CLINICAL TRIAL: NCT05404308
Title: Interest of a Weekly Consultation by a Medical Electro Radiology Manipulator (MERM) in Addition to the Follow-up by the Radiotherapist to Improve the Collection of Radio-induced Toxicities in Patients Undergoing Proton Therapy: Randomized Controlled Trial
Brief Title: Interest of a Weekly Consultation by a Medical Electro Radiology Manipulator (MERM) in Addition to the Follow-up by the Radiotherapist to Improve the Collection of Radio-induced Toxicities in Patients Undergoing Proton Therapy
Acronym: MERMOSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A00499-32
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Paramedical Consultation; Radiotherapy; Proton Therapy; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weekly follow-up by a medical radiography technician and weekly follow-up by the radiotherapist (Experimental)
  Interventions: Other: Consultation with Manipulator in Medical Radiology and a radiotherapist
- Standard weekly follow-up by the radiotherapist only (Active Comparator)
  Interventions: Other: Consultation with a radiotherapist

INTERVENTIONS:
Other: Consultation with Manipulator in Medical Radiology and a radiotherapist — Weekly consultation with Manipulator in Medical Radiology and a radiotherapist
  Arms: Weekly follow-up by a medical radiography technician and weekly follow-up by the radiotherapist
Other: Consultation with a radiotherapist — Weekly consultation with a radiotherapist
  Arms: Standard weekly follow-up by the radiotherapist only

SUMMARY:
To our knowledge, the investigators have not found any scientific article dealing with cooperation between radiation oncologists and medical radiation technologists in the context of monitoring patients undergoing radiotherapy. Cooperation protocols between health professionals are in progress but concern mainly technical procedures (ultrasound, laserthermal sessions).

This study aims to evaluate whether MERMs, after training by physicians, can monitor clinical signs (for usual well-described toxicities) during treatment via a dedicated consultation.

This approach participates in the development of new professions and cooperation protocols between health professionals. This mission of accompaniment on a dedicated time would make it possible to develop the caring role of the medical electroradiology manipulator.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years;
* Patient with malignant or benign brain or upper aerodigestive tract (ADT) tumor candidate for proton therapy;
* WHO score < 2
* Mastery of the French language;
* Patient affiliated with a social security system;
* Signature of informed consent prior to any specific procedure related to the study.

Exclusion Criteria:

* Patient with another cancer previously treated with radiation therapy;
* Simultaneous participation in a therapeutic clinical trial;
* Patient deprived of liberty or under guardianship;
* Any associated medical or psychological condition that may compromise the patient's ability to participate in the study
* Patient unable to undergo trial monitoring for geographical, social or psychopathological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with at least one toxicity requiring intervention | 3 weeks

SECONDARY OUTCOMES:
Number of toxicities detected | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No